CLINICAL TRIAL: NCT03427034
Title: Determining the Specificity and Sensitivity of the BladderLight™ Assay as a Diagnostic and Risk Stratification Tool for Bladder Cancer
Brief Title: Assessment of BladderLight SurvEILlance
Acronym: ABSEIL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Cytosystems Ltd (Unknown)
Responsible Party: Principal Investigator, Kasra Saeb-Parsy BSc, MB BS, AFHEA, FRCSEd (Urol), Consultant Urologist, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A094687
Record Dates: First submitted 2018-01-30; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Bladder Cancer
Keywords: Urine; Haematuria; Flexible cystoscopy; Recurrence; Cytology
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hematuria; Recurrence

STUDY DESIGN:
Intervention Model Description: all eligible patients will be recruited
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cystoscopic surveillance (Experimental): Patients with previous history of bladder cancer undergoing flexible cystoscopy will privide a urine sample to see if BladderLight system can exclude presence of bladder cancer
  Interventions: Device: BladderLight®
- Haematuria group (Experimental): Patients referred with haematuria to exclude bladder cancer will privide a urine sample to see if BladderLight system can exclude presence of bladder cancer
  Interventions: Device: BladderLight®
- Longitudinal group (No Intervention): Patient with Negative cystoscopy with a positive BladderLight® test will be followed for 12 months to see if they subsequently develop bladder cancer.

INTERVENTIONS:
Device: BladderLight® — Using a cell collection device to look for the presence of bladder cancer cells
  Arms: Cystoscopic surveillance; Haematuria group

SUMMARY:
Is BladderLight® (BL) urine testing accurate, as a non-invasive method, to exclude presence of bladder cancer in patients.

DETAILED DESCRIPTION:
There are three arms to the proposed performance evaluation of the integrated test - arms 1 and 2 are cross-sectional studies examining the accuracy of the BladderLight® test in the detection of cancer of the urinary bladder in patients attending either Gross Haematuria clinic for a potential primary (first time) diagnosis (arm 1) or patients attending Cystsoscopic Surveillance clinic as follow up to a previous, treated case of bladder cancer (arm 2). Arm 3 is a longitudinal examination of disease state following a negative cystoscopy with a positive BladderLight® test - this will examine whether BladderLight® can predict progression to overt disease. Arm three will not involve any further requirement for physical sampling, but will involve result checking on subsequent cystoscopies

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years of age or above.
2. Patients attending Cystoscopic Surveillance clinic for monitoring of recurrence of urothelial carcinoma after having been treated for urothelial carcinoma / bladder cancer (Arm 1) OR Patients attending Gross Haematuria clinic (or equivalent) for cystoscopy/biopsy (if appropriate) relating to symptoms suggestive of possible urothelial cancer (Arm 2). Patients that will receive a cystoscopy as per standard practice.
3. Able to understand and sign the written Informed Consent Form.
4. Able and willing to follow the Protocol requirements

Exclusion Criteria:

1. Participation in any clinical study of an Investigational Medicinal Product during the 8 weeks preceding the sampling period of the study.
2. Patients that have a urinary tract stent, kidney stones or catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
To exclude presence of bladder cancer with sensitivity of 85% | 12 month
  In each cohort of the study sensitivity, specificity, negative and positive predictive value for detection of cancer will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: kasra Saeb-Parsy, MBBS, FRCSEd, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Undecided
Data will be published in peer reviewed journals and presented at scientific meetings

REFERENCES:
- [Background] Saeb-Parsy K, Wilson A, Scarpini C, Corcoran M, Chilcott S, McKean M, Thottakam B, Rai B, Nabi G, Rana D, Perera M, Stewart K, Laskey RA, Neal DE, Coleman N. Diagnosis of bladder cancer by immunocytochemical detection of minichromosome maintenance protein-2 in cells retrieved from urine. Br J Cancer. 2012 Oct 9;107(8):1384-91. doi: 10.1038/bjc.2012.381. Epub 2012 Sep 11. PMID 22968648